CLINICAL TRIAL: NCT06787196
Title: Effect of Single Dose Intravenous Dexamethasone on Postoperative Pain and Complications in Jaw Surgery Under General Anesthesia
Brief Title: Intravenous Dexamethasone on Postoperative Pain and Complications in Jaw Surgery
Acronym: DXM-PAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, FUNDA ARUN, Assistant Professor Dr., Selcuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: F003
Record Dates: First submitted 2024-12-27; First posted 2025-01-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Tooth Extraction Status Nos; Cysts Dental; General Anesthesia
Keywords: Dexamethasone; postoperative pain; maxillofascial surgery
MeSH Terms: conditions — Radicular Cyst; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dexamethasone (Experimental): At the end of the procedure, patients received a single IV dose of Dexamethasone (0.1 mg/kg) before being extubated.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone, single-dose, 8 mg IV administered intraoperatively
  Other Names: Dekort

SUMMARY:
This study aims to evaluate the effect of single-dose intravenous dexamethasone on postoperative pain and other complications in compacted tooth and cyst enucleation procedures performed under general anesthesia.

DETAILED DESCRIPTION:
During surgery, patients were carefully monitored with standard equipment to track oxygen levels (SpO2), heart activity (ECG), blood pressure, and carbon dioxide levels. General anesthesia was started with medications like thiopental, rocuronium, and fentanyl, and maintained with a mix of oxygen, air, sevoflurane, and remifentanil. Patients were intubated with appropriate tubes, and the surgical team applied a local anesthetic (Articaine with Epinephrine) to the area before starting the procedure. After the surgery, patients were given dexamethasone (DXM) and pantoprazole intravenously, then safely extubated and sent to recovery. All patients were discharged on the same day.

Postoperative recovery was assessed using pain scores (VAS) and physical evaluations. Pain levels were categorized as mild, moderate, or severe, and an analgesic was provided if the score exceeded 3. Facial swelling was measured by comparing pre- and post-surgery facial landmarks, with swelling classified into grades based on the percentage of change. Mouth opening was evaluated with a caliper to check for trismus (jaw stiffness), with results grouped into normal, mild, moderate, or severe grades depending on the degree of restriction. Follow-ups were conducted by an independent clinician on postoperative days 1, 2, and 7.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* underwent split-mouth surgery

Exclusion Criteria:

* Patients undergoing corticosteroid therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
IV dexamethasone (DXM) changes postoperative complications | 6 months
  Postoperative pain, swelling, and restricted mouth opening are identified as key postoperative concerns. The anti-inflammatory effects of dexamethasone (DXM) are utilized to address these complications.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Kucukkolbasi, prof., Study Chair — Selcuk University; Emine Taskin, resid., Study Chair — Selcuk University
Locations (1):
- Funda Arun, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT06787196/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT06787196/ICF_001.pdf